CLINICAL TRIAL: NCT01281618
Title: Influence of Acid Reflux on Stromal Epithelial Interaction in Barrett's Esophagus
Acronym: CR20
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Prasad G. Iyer, MD, Mayo Clinic
Other Study IDs: 07-004899
Record Dates: First submitted 2011-01-20; First posted 2011-01-24 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2013-05

CONDITIONS: Barrett's Esophagus
Keywords: Barrett's esophagus
MeSH Terms: conditions — Barrett Esophagus | interventions — Gastroscopy; Endoscopy, Digestive System

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue specimens from Barrett's esophagus
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Those with barrett's esophagus: Those with barrett's esophagus: no dysplasia or low grade dysplasia
  Interventions: Procedure: 24 hour pH study and upper endoscopy (EGD)

INTERVENTIONS:
Procedure: 24 hour pH study and upper endoscopy (EGD) — All subjects enrolled will undergo 24 hour pH followed by EGD.

SUMMARY:
The purpose of this study is to determine the association between acid reflux and cell changes in Barrett's esophagus.

Specific aim 1: To test the hypothesis that controlled acid reflux is associated with lesser degree of stromal activation.

Specific aim 2: To test the hypothesis that stromal fibroblast derived growth factors drive BE epithelial proliferation.

ELIGIBILITY:
Inclusion Criteria:

1. Prior histological demonstration of Barrett's esophagus that is endoscopically visible; length of visible segment >/= 1 cm
2. Absence of dysplasia or LGD on biopsies within the past 5 years
3. Ability to provide informed consent
4. Age between 18 years and 90 years at study entry.

Exclusion criteria:

1. Eastern Cooperative Oncology Group performance status 3 or 4
2. Inability to tolerate endoscopic procedures
3. Pregnancy: Females of child-bearing age will be screened with pregnancy test.
4. Prior esophageal surgery, or cancer

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those diagnosed with barrett's esophagus confirmed by pathology with no dysplasia or low grade dysplasia
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2008-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
activated myofibroblasts | 6 months
  The primary end point for the study will be the proportion of patients with activated myofibroblasts (defined as positive staining for SMA and vimentin with negative staining for Desmin, in > 50% of subepithelial myofibroblasts). This primary end point will be compared between the group with controlled acid reflux and the group without acid reflux.

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States